CLINICAL TRIAL: NCT03215589
Title: A Prospective Study of Cerebral Oximetry to Assess Symmetry of Cerebral Blood Flow and Clinical Outcomes in Cardiac Surgery Patients Undergoing Hypothermic Circulatory Arrest
Brief Title: Assessment of Cerebral Blood Flow Asymmetry in Cardiac Surgery Patients Undergoing Hypothermic Circulatory Arrest
Acronym: COASTLINE
Status: Terminated | Type: Observational
Why Stopped: due to a change in surgical personnel, the operative technique changed, precluding the examination of bypass-related bi-hemispheric saturation differences.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2017:002
Record Dates: First submitted 2017-07-04; First posted 2017-07-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2018-06

CONDITIONS: Cerebral Desaturation; Cerebral Ischemia
Keywords: Near-infrared spectroscopy-derived cerebral oximetry
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral oxygen desaturation during cardiac surgery measured using near infrared spectroscopy (NIRS) derived cerebral oximetry has been associated with significant postoperative morbidity. If significant desaturation occurs during this period, it may represent an ideal opportunity to further optimize the postoperative care of these patients.

DETAILED DESCRIPTION:
Selective antegrade cerebral perfusion (SACP) is a commonly used technique for maintaining cerebral blood flow (CBF) during the use of hypothermic cardiac arrest (HCA) for aortic arch reconstruction. However, even with an intact Circle of Willis, asymmetric CBF is a common occurrence during HCA when SACP is used. The investigators have previously shown that ultrasound guided extrinsic compression of the left carotid artery can increase left cerebral oxygen saturation, and improved symmetry of CBF; however, this has not been investigated formally. In this study, the investigators will firstly formally assess the incidence and severity of asymmetrical cerebral flow between the left and right hemispheres in patients undergoing aortic arch repair (n=20). CBF will be assessed indirectly through regional cerebral oxygen saturation (rSO2) measured via near-infrared spectroscopy-derived cerebral oximetry. In addition, a number of clinical outcome parameters (up to 30 days post-op) will be evaluated. The investigators expect that significant left-side cerebral hypoperfusion will consistently be observed in patients undergoing aortic arch repair using SACP.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18 years or older
* Surgery requiring cardio pulmonary bypass
* Ascending aorta or arch repair surgery
* Surgery requiring hypothermic circulatory arrest

Exclusion Criteria:

* Off-pump cardiac surgery
* Skin condition preventing the use of cerebral oximetry pads

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 20 consecutive patients undergoing cardiac surgery employing CPB will be studied
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of asymmetrical cerebral desaturation | Duration of hypothermic circulatory arrest between surgical induction and ICU admission
  Cerebral desaturation defined as a greater than 10% difference in cerebral saturation comparing one hemisphere to the other based on a baseline reading taken in the minute preceding the onset of HCA to the end of the hypothermic period.

SECONDARY OUTCOMES:
Severity of asymmetrical cerebral desaturation | Duration of hypothermic circulatory arrest between surgical induction and ICU admission
  Area of the curve (AUC) and time under the curve (TUC) for all saturation events less than pre-induction baseline as well as for 10%, 15% and 25%, relative reductions under the baseline rSO2 will also be determined. In addition, the AUC and TUC for rSO2 less than an absolute rSO2 of 50% will also be determined.
Severity of asymmetrical cerebral desaturation | Duration of hypothermic circulatory arrest between surgical induction and ICU admission
  Time under the curve (TUC) for all saturation events less than pre-induction baseline as well as for 10%, 15% and 25%, relative reductions under the baseline rSO2 will also be determined. In addition, the AUC and TUC for rSO2 less than an absolute rSO2 of 50% will also be determined.
All cause mortality | Surgical induction to 30 day postoperative
  All cause mortality
Neurologic injury | Surgical induction to 30 day postoperative
  Any neurologic injury, including: stroke, delirium, seizures, coma
Renal injury | Surgical induction to 30 day postoperative
  Renal injury defined as a 50% decrease in estimated glomerular filtration rate (GFR) and/or need for dialysis
Serious infection | Surgical induction to 30 day postoperative
  Serious infection including: mediastinitis, cellulitis, pneumonia, urinary tract infection
Gastrointestinal morbidity | Surgical induction to 30 day postoperative
  Gastrointestinal (GI) morbidity defined as GI bleed, bowel perforation and/or ischemia
In-hospital mortality | Surgical induction to hospital discharge or 30 days postoperative, whichever comes first
  In hospital mortality
Hospital length of stay | Surgical induction to hospital discharge or 30 days postoperative, whichever comes first
  The length of time (in days) that the patient remained in the hospital after surgery
ICU length of stay | ICU admission to ICU discharge or 30 days postoperative, whichever comes first
  length of stay in the intensive care unit
Intubation time | Time of surgical intubation to time of extubation
  Duration of time that the patient was intubation from the start of surgery
Transfusions | Surgical induction to hospital discharge or 30 days postoperative, whichever comes first
  The need for transfusions, including: red blood cells, platelets, plasma and cryoprecipitate
Renal function | Preoperative to hospital discharge or 30 days postoperative, whichever comes first
  Greatest percent change in creatinine and 25% and 50% increase in creatinine
Hemostatic support | ICU admission to hospital discharge or 30 days postoperative, whichever comes first
  Requirement of vasopressors, intra-aortic balloon pumps (IABPs) and inotropes (0-12 hours, 12-24 hours and >24 hours post-operative
Atrial fibrillation | ICU admission to hospital discharge or 30 days postoperative, whichever comes first
  Atrial fibrillation
Myocardial infarction | ICU admission to hospital discharge or 30 days postoperative, whichever comes first
  Myocardial infarction as defined by:
Atrial and/or ventricular arrhythmia | ICU admission to hospital discharge or 30 days postoperative, whichever comes first
  Atrial and/or ventricular arrhythmia, requiring electrical or pharmacologic intervention
Nausea and vomiting | ICU admission to hospital discharge or 30 days postoperative, whichever comes first
  Excess nausea and vomiting, requiring more than one drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hilary P Grocott, MD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Fischer GW, Lin HM, Krol M, Galati MF, Di Luozzo G, Griepp RB, Reich DL. Noninvasive cerebral oxygenation may predict outcome in patients undergoing aortic arch surgery. J Thorac Cardiovasc Surg. 2011 Mar;141(3):815-21. doi: 10.1016/j.jtcvs.2010.05.017. Epub 2010 Jun 25. PMID 20579669